CLINICAL TRIAL: NCT00236847
Title: Double-Blind, Parallel Comparison of Topiramate 300 mg Twice Daily to Placebo in Patients With Refractory Partial Epilepsy
Brief Title: A Study of the Efficacy and Safety of Topiramate in the Treatment of Patients With Epilepsy.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR005566
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-04

CONDITIONS: Epilepsy; Epilepsies, Partial; Seizures
Keywords: topiramate; epilepsy; partial epilepsy; seizures; epileptic seizures; partial seizure disorder; brain diseases
MeSH Terms: conditions — Epilepsy; Epilepsies, Partial; Seizures; Brain Diseases | interventions — Topiramate

INTERVENTIONS:
Drug: topiramate

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of topiramate as an add-on therapy in patients with uncontrolled partial onset seizures who are taking one or two standard antiepileptic drugs.

DETAILED DESCRIPTION:
Epilepsy is characterized by seizures, which are abnormal electrical discharges in the brain that temporarily disrupt normal brain function. Seizures are classified as "generalized," originating in both sides of the brain simultaneously, or "partial-onset," starting in one area of the brain. Antiepilepsy medications, such as topiramate, are selected based on seizure type. This study is designed to study patients with partial epilepsy. This is a double-blind, placebo-controlled study that includes a baseline phase and a treatment phase. During the baseline phase (8 weeks duration), patients receive one or two standard antiepileptic drugs (AEDs), such as phenytoin, carbamazepine, phenobarbital, primidone, or valproic acid. Patients who continue to have seizures during treatment with standard AEDs proceed into the double-blind treatment phase. Patients then receive topiramate or placebo at a dosage of 100-milligrams (mg) once daily, increasing gradually to 3 tablets twice daily (600 mg/day, maximum) for 12 weeks (total duration of double-blind phase), while continuing on their standard AED regimen. Assessments of effectiveness include the percent reduction in the average monthly seizure rate, percent of patients responding to treatment (having equal to or greater than 50% reduction in seizure rate), and the patient's and investigator's global assessments of medication at end of study. Safety assessments include the incidence of adverse events throughout the study, clinical laboratory tests (hematology, serum chemistry, urinalysis), neurologic examinations, and vital sign measurements (blood pressure, pulse, temperature) weekly during the treatment phase. The study hypothesis is that topiramate, taken as add-on therapy to treatment with AEDs, will significantly reduce seizure frequency, compared with placebo, in patients with refractory partial epilepsy: that is, in patients who continue to have seizures despite treatment with a first-line AEDs. In addition, it is hypothesized that topiramate is well-tolerated. Topiramate, 100 milligrams (mg) oral tablets. Dosage begins at 100 mg once daily and increases gradually over 4 weeks to 3 tablets twice daily (600 mg/day, maximum) or maximum tolerated dose for an additional 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* History of simple or complex partial epilepsy that has been documented or witnessed
* an electroencephalogram (EEG) during the preceding 5 years that has a pattern consistent with the diagnosis of partial epilepsy
* during an 8-week baseline phase, patient must have at least 8 partial seizures while maintaining therapeutic levels of antiepileptic drugs (AEDs) and have no more than one seizure-free interval of up to 3 weeks
* and no seizure-free interval longer than 3 weeks
* good physical health.

Exclusion Criteria:

* Patients having solely generalized seizures or lacking documentation of partial epilepsy
* patients with generalized tonic-clonic seizures or other generalized epilepsies in the absence of an EEG consistent with partial epilepsy
* generalized seizures, which are defined by the EEG wave pattern
* seizures that lack an abnormal pulsation pattern on EEG
* females who are pregnant, nursing, or those not using adequate birth control if capable of having children

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 1989-12; Study Completion 1993-07 (Actual)

PRIMARY OUTCOMES:
Percent reduction in the average monthly seizure rate from baseline to end of treatment

SECONDARY OUTCOMES:
Percent of patients responding to treatment (>= 50% reduction in seizure rate from baseline to end of treatment); patient's and investigator's global assessments at end of study; incidence of adverse events throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Tassinari CA, Michelucci R, Chauvel P, Chodkiewicz J, Shorvon S, Henriksen O, Dam M, Reife R, Pledger G, Karim R. Double-blind, placebo-controlled trial of topiramate (600 mg daily) for the treatment of refractory partial epilepsy. Epilepsia. 1996 Aug;37(8):763-8. doi: 10.1111/j.1528-1157.1996.tb00649.x. PMID 8764816
- See also: A study of the efficacy and safety of topiramate in the treatment of patients with epilepsy — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=666&filename=CR005566_CSR.pdf